CLINICAL TRIAL: NCT05930730
Title: A Phase 2, Non-inferiority, Open-label, Randomized Controlled Study to Evaluate the Immunogenicity and Safety of Comvigen (Bivalent) Vaccine as a Booster Dose in Adults Who Have Received a Previous Booster Dose of an Approved COVID-19 Vaccine
Brief Title: Immunogenicity and Safety of Comvigen (Bivalent) Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Chula Clinical Research Center (Chula CRC), Faculty of Medicine Chulalongkorn University, Bangkok, Thailand (Unknown); HIV-NAT, Thai Red Cross - AIDS Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ChulaVac 006
Record Dates: First submitted 2023-06-20; First posted 2023-07-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Safety of a Single Dose of COMVIGEN Vaccine; Reactogenicity of a Single Dose of COMVIGEN Vaccine; Immunogenicity of a Single Dose of COMVIGEN Vaccine; Safety of a Single Dose of BIVALENT Pfizer/BNT Vaccine; Reactogenicity of a Single Dose of BIVALENT Pfizer/BNT Vaccine; Immunogenicity of a Single Dose of BIVALENT Pfizer/BNT Vaccine
Keywords: Non-inferiority study; Open-label; Randomized Controlled Study; Immunogenicity of the booster dose; safety of booster dose; reactogenicity of booster dose; COMVIGEN (Bivalent, ChulaCov19 BNA159.2 vaccine); Pfizer bivalent vaccine (Comirnaty, BIVALENT); mRNA from the ancestral (original) strain; Omicron variant (BA.4/BA.5) of SARS-CoV-2
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comvigen (Bivalent, ChulaCov19 BNA159.2) (Experimental)
  Interventions: Biological: Comvigen (Bivalent, ChulaCov19 BNA159.2)
- BIVALENT Pfizer/BNT vaccine (Active Comparator)
  Interventions: Biological: BIVALENT Pfizer/BNT vaccine

INTERVENTIONS:
Biological: Comvigen (Bivalent, ChulaCov19 BNA159.2) — single dose of COMVIGEN at 50 ug, as a booster dose, given at 3 months and above after receipt of a previous booster dose of any approved mRNA COVID-19 vaccine
  Arms: Comvigen (Bivalent, ChulaCov19 BNA159.2)
Biological: BIVALENT Pfizer/BNT vaccine — single dose of BIVALENT of Pfizer/BNT Bivalent vaccine at 30 ug, as a booster dose, given at 3 months and above after receipt of a previous booster dose of any approved mRNA COVID-19 vaccine
  Arms: BIVALENT Pfizer/BNT vaccine

SUMMARY:
This study will assess the safety, reactogenicity and immunogenicity of a single dose of Comvigen (Bivalent, ChulaCov19 BNA159.2) vaccine or BIVALENT Pfizer/BNT vaccine as a booster among healthy males and non-pregnant females aged 18-64 years after receiving a previous booster dose of any approved mRNA COVID-19 vaccine for more than 3 months. The results of Combiven will be compared to BIVALENT Pfizer/BNT vaccine.

DETAILED DESCRIPTION:
This is a phase II, non-inferiority, multicenter randomized open-label trial in which 450 healthy males and non-pregnant females, aged 18-64 years, will be recruited from multi-sites in Thailand. The randomization will be a 2:1 design to receive either Comvigen (Bivalent, ChulaCov19 BNA159.2) vaccine or BIVALENT Pfizer/BNT vaccine. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of a single dose of COMVIGEN at 50 ug, as a booster dose, given at 3 months and above after receipt of a previous booster dose of any approved mRNA COVID-19 vaccine. The estimated sample size would also allow a comparison between a booster dose, Comvigen (Bivalent, ChulaCov19 BNA159.2) vaccine at 50 ug to Comirnaty, BIVALENT of Pfizer/BNT Bivalent vaccine at 30 ug dose.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all the following criteria at Screening are eligible to participate in the study:

1. Must be a male or female aged 18 - 64 (inclusive) at the time of enrolment
2. Must have completed at least a primary course of 2 doses of any approved COVID-19 vaccine which the last dose have to be mRNA vaccine and completed the last doser 3 months or more
3. Must be able to communicate effectively with study personnel and considered reliable, willing, and cooperative in terms of compliance with the protocol requirements
4. Participants must sign the written informed consent form prior to undertaking any protocol-related procedures
5. SARS-CoV-2 rapid antigen test is negative at Day 1 (the day of receiving the study booster dose)
6. Does not intend to receive any other authorized/approved COVID-19 vaccine at the time of enrolment and up to 3 months of the study
7. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), practice true abstinence or, if engaged in sexual relations with a female of child-bearing potential, the participants and their partner must use an acceptable, highly effective, double-barrier contraceptive method* from Screening and for a period of at least 60 days after vaccination
8. A female participant is eligible if she is not pregnant, or breastfeeding indicated by one of the following conditions:

   1. With childbearing potential (WOCBP): she agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to the study intervention administration until at least 12 weeks after the study intervention administration, or
   2. With non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile
9. Participants must be in general good health* based on medical history and physical examination, as determined by the PI at Screening.
10. Participants must agree to refrain from donating blood, plasma, ova, sperm, or organs during the whole study.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible to participate in the study:

1. History of a systemic hypersensitivity or life-threatening reaction to a vaccine containing any of the same or similar substances.
2. History of test-confirmed by PCR or rapid antigen test to SARS-CoV-2 COVID-19 infection within 3 months prior to randomisation.
3. Presence of clinically significant medical history*, unstable chronic or acute disease that, in the opinion of the PI, may increase the risk of exposure to the investigational vaccine
4. History of having any significant side effects after receipt of any other COVID-19 vaccine eg. endocarditis, pericarditis or myocarditis. History of any severe reactogenic side effects or other medical illness that were thought to be associated with vaccine.
5. Presence of an acute illness* or with fever at 38.00 C or more within 72 hours prior to vaccination.
6. Bleeding disorders or taking an anticoagulant or anti-platelet agent that may contraindicate for intramuscular injection based on Investigator's judgment
7. Inadequate venous access to allow the collection of blood samples.
8. Received any prophylactic or therapeutic vaccine, biologic product, device or blood product, within 4 weeks of vaccination or 5 half-lives (whichever is longer) or anticipate doing so in the follow-up period defined for this study. For influenza vaccine, however, can be administered up to 14 days prior to randomization and following visit 3 (Day 29+3) after blood sample collection.
9. History of ever had an anaphylaxis reaction to food, medication, or vaccination.
10. Participant is immunosuppressed as caused by disease or immunosuppressive therapy or anticipated need to use of any chemotherapy or immunosuppressive agents* within the next 6 months.
11. Participation in any of the other investigational trials of vaccines, therapeutic, or medical devices 12 weeks before or during the 6 months of this study.
12. Received immunoglobulins and/or any blood or blood products within 3 months before vaccination day or plans to receive any blood or blood products at any time during the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
adverse events | 30 minutes after vaccination
  Presence of immediate adverse events within 30 minutes after vaccination
solicited injection site or systemic reactions | within 7 days after vaccination
  Presence of solicited injection site or systemic reactions within 7 days after vaccination
unsolicited adverse events | within 28 days after vaccination
  Presence of unsolicited adverse events within 28 days after vaccination
serious adverse events (SAEs) | 169 days
  Presence of serious adverse events (SAEs) from day 1 to Day 169
medically attended adverse events (MAAEs) | 169 days
  Presence of medically attended adverse events (MAAEs) from day 1 to Day 169
New Onset Chronic Medical Condition (NOCMCs) | 169 days
  Presence of New Onset Chronic Medical Condition (NOCMCs) from day 1 to Day 169
vital signs | 169 days
  Number of participants with abnormal vital signs
vital signs | 169 days
  Percent of participants with abnormal vital signs
clinical changes | 169 days
  Number of participants with abnormal physical examinations finding
clinical changes | 169 days
  Percent of participants with abnormal physical examinations findingexaminations
Geometric mean titers of neutralizing antibody titer | Day 29
  Geometric mean titers of neutralizing antibody titer measured by pseudoviral neutralization assay (psVNT-50) against Omicron BA.4/BA.5 exposed to COMVIGEN (Bivalent) vaccine
Geometric mean titers of neutralizing antibody titer | Day 29
  Geometric mean titers of neutralizing antibody titer measured by pseudoviral neutralization assay (psVNT-50) against wild-type virus exposed to COMVIGEN (Bivalent) vaccine
Geometric mean titers of neutralizing antibody titer | Day 29
  Geometric mean titers of neutralizing antibody titer measured by pseudoviral neutralization assay (psVNT-50) against Omicron BA.4/BA.5 exposed to BIVALENT vaccine
Geometric mean titers of neutralizing antibody titer | Day 29
  Geometric mean titers of neutralizing antibody titer measured by pseudoviral neutralization assay (psVNT-50) against wild-type virus exposed to BIVALENT vaccine
Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer | Day 29
  Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer against wild-type virus exposed to COMVIGEN (Bivalent) vaccine
Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer | Day 29
  Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer against Omicron BA.4/BA.5 exposed to COMVIGEN (Bivalent) vaccine
Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer | Day 29
  Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer against wild-type virus exposed to BIVALENT vaccine
Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer | Day 29
  Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer against Omicron BA.4/BA.5 exposed to BIVALENT vaccine
Proportion of participants with at least 4-fold-rise in neutralizing antibody titer | Day 29
  Proportion of participants with at least 4-fold-rise in neutralizing antibody titer, psVNT-50 against wild-type virus exposed to COMVIGEN (Bivalent)
Proportion of participants with at least 4-fold-rise in neutralizing antibody titer | Day 29
  Proportion of participants with at least 4-fold-rise in neutralizing antibody titer, psVNT-50 against Omicron BA.4/BA.5 exposed to COMVIGEN (Bivalent)
Proportion of participants with at least 4-fold-rise in neutralizing antibody titer | Day 29
  Proportion of participants with at least 4-fold-rise in neutralizing antibody titer, psVNT-50 against against wild-type virus exposed to BIVALENT vaccine
Proportion of participants with at least 4-fold-rise in neutralizing antibody titer | Day 29
  Proportion of participants with at least 4-fold-rise in neutralizing antibody titer, psVNT-50 against against Omicron BA.4/BA.5 exposed to BIVALENT vaccine

SECONDARY OUTCOMES:
Geometric mean titers of neutralizing antibody titer | Day 29
  Geometric mean titers of neutralizing antibody titer at Day 29 measured by psVNT-50 against other relevant variants of concerns (VOCs)
Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer | Day 29
  Geometric mean of the fold-rise post-vaccination of psVNT-50 neutralizing antibody titer against other relevant VOCs from Day 1 to Day 29
Proportion of participants with at least 4-fold-rise in neutralization antibody titer | Day 29
  Proportion of participants with at least 4-fold-rise in neutralization antibody titer, psVNT-50 against other relevant VOCs from Day 1 to Day 29
Geometric mean titers of neutralizing antibody titer | Day 1
  Geometric mean titers of neutralizing antibody titer at Day 1 measured by live-virus microneutralization assay (micro-VNT-50) against wild-type virus
Geometric mean titers of neutralizing antibody titer | Day 29
  Geometric mean titers of neutralizing antibody titer at Day 29 measured by live-virus microneutralization assay (micro-VNT-50) against wild-type virus
Geometric mean titers of neutralizing antibody titer | Day 1
  Geometric mean titers of neutralizing antibody titer at Day 1 measured by live-virus microneutralization assay (micro-VNT-50) against omicron BA.4/BA.5
Geometric mean titers of neutralizing antibody titer | Day 29
  Geometric mean titers of neutralizing antibody titer at Day 29 measured by live-virus microneutralization assay (micro-VNT-50) against omicron BA.4/BA.5
Geometric mean of the fold-rise post-vaccination of micro-VNT-50 | Day 29
  Geometric mean of the fold-rise post-vaccination of micro-VNT-50 against wild-type on Day 29.
Geometric mean of the fold-rise post-vaccination of micro-VNT-50 | Day 29
  Geometric mean of the fold-rise post-vaccination of micro-VNT-50 against omicron BA.4/BA.5 virus on Day 29.
Proportion of participants with at least 4-fold-rise in micro-VNT-50 | Day 29
  Proportion of participants with at least 4-fold-rise in micro-VNT-50 against wild-type virus on Day 29.
Proportion of participants with at least 4-fold-rise in micro-VNT-50 | Day 29
  Proportion of participants with at least 4-fold-rise in micro-VNT-50 against omicron BA.4/BA.5 virus on Day 29.
Geometric mean titers of anti-RBD antibody titer | Day 29
  Geometric mean titers of anti-RBD antibody titer at Day 29 against wild type.
Geometric mean titers of anti-Spike (S) antibody titer | Day 29
  Geometric mean titers of anti-Spike (S) antibody titer at Day 29 against wild type.
Geometric mean of the fold-rise post-vaccination of anti-RBD antibody | Day 29
  Geometric mean of the fold-rise post-vaccination of anti-RBD antibody against wild-type virus at Day 29.
Geometric mean of the fold-rise post-vaccination of anti-S antibody titer | Day 29
  Geometric mean of the fold-rise post-vaccination of anti-S antibody titer against wild-type virus at Day 29.
Proportion of participants with at least 4-fold-rise in anti-RBD | Day 29
  Proportion of participants with at least 4-fold-rise in anti-RBD titer against wild-type virus at Day 29
Proportion of participants with at least 4-fold-rise in anti-RBD | Day 29
  Proportion of participants with at least 4-fold-rise in anti-S antibody titer against wild-type virus at Day 29
Geometric mean of SARS-CoV2-specific T-cell responses | Day 1
  Geometric mean of SARS-CoV2-specific T-cell responses (spot-forming cells or SFC per 1 million PBMCs) measured by IFN gamma-ELISPOT assay against wild-type peptides at day 1
Geometric mean of SARS-CoV2-specific T-cell responses | Day 29
  Geometric mean of SARS-CoV2-specific T-cell responses (spot-forming cells or SFC per 1 million PBMCs) measured by IFN gamma-ELISPOT assay against wild-type peptides at day 29
median number of SARS-CoV2-specific T-cell responses | Day 1
  median number of SARS-CoV2-specific T-cell responses (spot-forming cells or SFC per 1 million PBMCs) measured by IFN gamma-ELISPOT assay against wild-type peptides at day 1
median number of SARS-CoV2-specific T-cell responses | Day 29
  median number of SARS-CoV2-specific T-cell responses (spot-forming cells or SFC per 1 million PBMCs) measured by IFN gamma -ELISPOT assay against wild-type peptides at day 29
Geometric mean of the fold-rise post-vaccination of SARS-CoV2-specific T-cell responses | Day 29
  Geometric mean of the fold-rise post-vaccination of SARS-CoV2-specific T-cell responses (spot-forming cells (SFC) per 1 million PBMCs) measured by IFN gamma-ELISPOT assay against wild-type peptides exposed to COMVIGEN (Bivalent) vaccine on Day 29
Geometric mean of the fold-rise post-vaccination of SARS-CoV2-specific T-cell responses | Day 29
  Geometric mean of the fold-rise post-vaccination of SARS-CoV2-specific T-cell responses (spot-forming cells (SFC) per 1 million PBMCs) measured by IFN gamma-ELISPOT assay against wild-type peptides exposed to BIVALENT vaccine on Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Watsamon Jantarabenjakul, MD, Principal Investigator — Department of Pediatric, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand; Sivaporn Gatechompol, MD, Principal Investigator — HIVNAT, Thai Red Cross AIDS Research Centre, Bangkok, Thailand
Locations (2):
- Thailand (2):
  - Department of Pediatric, Faculty of Medicine, Chulalongkorn University, Bangkok
  - HIV-NAT, Thai Red Cross - AIDS Research Centre, Bangkok

REFERENCES:
- [Derived] Jantarabenjakul W, Nantanee R, Puthanakit T, Gatechompol S, Avihingsanon A, Punrin S, Tantawichien T, Nitayaphan S, Thitithanyanont A, Buranapraditkun S, Jongkaewwattana A, Ketloy C, Prompetchara E, Lawpoolsri S, Wijagkanalan W, Alameh MG, Hong L, Samija M, Weissman D, Ruxrungtham K; ChulaVac006 Study Team. Immunogenicity and safety of 'Comvigen', a bivalent SARS-CoV-2 vaccine, in comparison to Comirnaty bivalent vaccine in Thailand: a phase 2, non-inferiority randomised trial. Lancet Reg Health Southeast Asia. 2025 Aug 15;40:100650. doi: 10.1016/j.lansea.2025.100650. eCollection 2025 Sep. PMID 40895389